CLINICAL TRIAL: NCT04389099
Title: MRI Angiography of Physiological and Pathological Pregnancy Placentas Ex-vivo
Acronym: MAPLE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BERTHOLDT Charline, Principal Investigator (gynecologist-obstetrician), Central Hospital, Nancy, France
Other Study IDs: PSS2018/MAPLE-BERTHOLDT/SKJ
Record Dates: First submitted 2020-05-06; First posted 2020-05-15 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pre-Eclampsia; Fetal Growth Retardation
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy placenta (control): Pregnant women without preeclampsia and/or fetal growth restriction
- Pathological placenta: Pregnant women with preeclampsia and/or fetal growth restriction divided into two subgroups : preeclampsia with or without fetal growth restriction ; fetal growth restriction without preeclampsia.

SUMMARY:
Introduction:

The placenta is the organ that permits the maternal-fetal exchange of the oxygen and nutrients. The development of its vascular network occurs in the first trimester. Any deficit during this important angiogenesis procedure can lead to the dysfunction of the placental vasculature, which can potentially cause pathologies including preeclampsia (PE) and intrauterine growth restriction (IUGR). PE concerns 3% of the pregnancy in France. It can occur at any gestational age and leads to serious complications such as eclampsia, the HELLP syndrome or the retro-placental hematoma. IUGR does not only lead to the morbidity and fetal and neonatal mortality, but also has a predisposition for certain pathologies in the adulthood.

Many groups have studied the placenta vasculature at the microscopic (histological) scale. However, recent studies show that in addition to the damage at the microvasculature level, the macroscopic placental vessel architecture is also altered. Nonetheless, the origin and the etiology of this phenomenon remains unknown.

Since it is difficult to apply in-vivo imaging techniques on pregnant women due to the restriction of usage of contrast agent. Alternatively, ex-vivo MR angiography (MRA) techniques have been developed by our team and others to visualize the entire placental vasculature in a faster way (as compared to corrosion casting). Up to now, only the study of the healthy placenta is done and published. The analysis of the pathological placental vasculature (i.e. PE and IUGR cases) at different gestational age and its comparison to the physiological ones have not been conducted, which will potentially enable a better understanding of the placental vasculature pathology.

Objectives: the main objective of this study is to compare the vasculature architecture of the normal and pathological placentas (with possible alteration in the placental vasculature).

Methods and analysis: This is a monocentric, prospective, controlled but not randomized study. The investigators expect to include 110 women in Nancy. The pregnant women will be recruited when they arrived at the maternity hospital for delivery, for both the physiological and potential pathological cases. The notice of this study will be given. If no opposition is given by the subject, the placenta may be collected. This study will not collect the patient consent but only the opposition declaration will be collected.

ELIGIBILITY:
Inclusion Criteria:

* already received the complete information about the study and do not express any opposition to the utilisation of their data
* mandatory enrolment in a social security plan
* gestational age more than 30 weeks (and until at term)
* patient with either natural delivery or with cesarean section and whose placenta is naturally completely separated (directed delivery only)

Exclusion Criteria:

* younger than 18 years old
* new borns with congenital disease (either suspected at birth or already diagnosed)
* presence of only one umbilical artery
* presence of a maternal pathology: gestational or pre-existing diabetes, autoimmune diseases that may have an impact on placental vascularization (Antiphospholipid Antibody Syndrome, Immune Thrombocytopenia, Myasthenia, Systemic Lupus Erythematosus), cancer,
* do not speak the French language, or inability to understand the given information of the study
* manual delivery
* incomplete placenta
* placenta with true marginal insertions (cord insertion within 1 cm of the placental margin) and/or velaments of the cord
* Person referred to Articles L.1121-6 and L-1121-8 of the Public Health Code

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * healthy placenta group: 50 inclusion (among which, 10 is to establish the final technical protocol)
  * pathological placenta group: 60 (30 preeclampsia and 30 intrauterine restricted growth only cases)
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2024-11-17 (Actual)

PRIMARY OUTCOMES:
Placental vasculature architecture indice: total vascular density | through study completion, on average of 24 months
Placental vasculature architecture indice: placental artery density (cm3) | through study completion, on average of 24 months
Placental vasculature architecture indice: placental vien density (cm3) | through study completion, on average of 24 months
Placental vasculature architecture indice: placental vessel tortuosity | through study completion, on average of 24 months
Placental vasculature architecture indice: placental vessel tree branching | through study completion, on average of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Charline BERTHOLDT, Study Chair — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Dap M, Chen B, Banasiak C, Hossu G, Morel O, Beaumont M, Bertholdt C. Magnetic Resonance Imaging Angiography of Physiological and Pathological Pregnancy Placentas Ex Vivo: Protocol for a Prospective Pilot Study. JMIR Res Protoc. 2022 Aug 10;11(8):e35051. doi: 10.2196/35051. PMID 35947435